CLINICAL TRIAL: NCT05474027
Title: Does Tranexamic Acid Reduce the Need for Deliberate Hypotensive Anesthesia Within Orthognathic Surgery? a Prospective Study
Brief Title: Reducing Hypotensive Anesthesia Use with TXA During Orthognathic Surgery
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Brian Kinard, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-300009440
Record Dates: First submitted 2022-07-20; First posted 2022-07-26 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Hypotension During Surgery; Blood Loss, Surgical
Keywords: orthognathic surgery
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Tranexamic Acid; Injections, Intravenous; Solutions

STUDY DESIGN:
Intervention Model Description: Our goal is to enroll 50 patients. Patients will be recruited from Dr. Kinard's regularly scheduled orthognathic cases at UAB Highlands Hospital. The patient will be informed of the study in advance and have consent signed pre-operatively. 1g of tranexamic acid will be given perioperatively as already routinely performed. The anesthesia team will be asked to avoid deliberate hypotensive anesthesia and maintain blood pressure closer to patient baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients Receiving Tranexamic Acid with Avoidance of Hypotensive Anesthesia (Experimental)
  Interventions: Other: Avoidance of Deliberate Hypotensive Anesthesia; Drug: TRANEXAMIC ACID 1 G in 10 mL INTRAVENOUS INJECTION, SOLUTION

INTERVENTIONS:
Other: Avoidance of Deliberate Hypotensive Anesthesia — The anesthesia team will be asked to avoid deliberate hypotensive anesthesia and maintain blood pressure closer to the patient's baseline throughout the surgery.
Drug: TRANEXAMIC ACID 1 G in 10 mL INTRAVENOUS INJECTION, SOLUTION — 1g of tranexamic acid will be given intravenously to patient undergoing orthognathic surgery as routinely performed about 5-15 minutes before first surgical incision.

SUMMARY:
This prospective study will analyze the need for deliberate hypotensive anesthesia (DHA) during orthognathic surgery when tranexamic acid (TXA) is administered. DHA has been proven to be effective although it comes with multiple risks related to organ hypoperfusion including kidney injury, stroke, and cardiac ischemia. Therefore, it may be potentially safer for patients to avoid deliberate hypotensive anesthesia if TXA alone adequately controls blood loss and provides adequate surgical site visualization.

DETAILED DESCRIPTION:
Our goal is to enroll 50 patients. Patients will be recruited from Dr. Kinard's regularly scheduled orthognathic cases at UAB Highlands Hospital. The patient will be informed of the study in advance and have consent signed pre-operatively. Patients will be evaluated for the following variables: sex, age, weight at time of surgery, preoperative hemoglobin, and preoperative hematocrit. Patients will be included if they are undergoing bimaxillary orthognathic surgery at UAB Highlands Hospital. All patients treated with orthognathic surgery already are provided 1g of TXA perioperatively and this will be continued through this study. All patients will be treated with 1g of TXA perioperatively and the anesthesia team will be instructed to limit deliberate hypotensive anesthesia unless otherwise directed by the surgeon. Perioperative and post-operative measurements will include: estimated blood loss, pre and post-operative hemoglobin, pre and post-operative hematocrit, average mean arterial pressure throughout the case (MAP), maximum MAP (excluding induction and emergence), minimum MAP (excluding induction and emergence), total MAP time under 65 mmHg, length of procedure, and surgeon evaluation of visual field throughout the procedure utilizing Fromme's ordinal scale. Based on these factors, it will help determine the need for deliberate hypotensive anesthesia during orthognathic surgery when tranexamic acid is administered.

ELIGIBILITY:
Inclusion Criteria:

* Bimaxillary orthognathic surgery completed at UAB Highlands Hospital

Exclusion Criteria:

* History of hypertension or previously diagnosed cardiac problems
* Bleeding diathesis
* TXA medically contraindicated

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Surgeon's Analysis of Surgical Field Visualization | 1 year
  The surgeon will evaluate surgical field visibility using Fromme's ordinal scale
Mean Arterial Pressure | 1 year
  Tracking mean arterial pressures throughout surgery, evaluating if patient's blood pressure can be reliably kept around patient's baseline instead of deliberate hypotensive anesthesia.
Estimated Blood Loss | 1 year
  Volume of blood loss recorded during surgical case

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kinard, DMD, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Hospital-Highlands, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No